CLINICAL TRIAL: NCT00839566
Title: Permanent Atrial Fibrillation in Heart Failure Trial
Brief Title: PAF-HEFT (Permanent Atrial Fibrillation in Heart Failure Trial)
Acronym: PAF-HEFT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Number of eligible patients too small.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_9
Record Dates: First submitted 2009-01-13; First posted 2009-02-09 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AV ablation (Experimental)
  Interventions: Procedure: Ablation
- Rate control (Active Comparator): Rate control by drugs
  Interventions: Other: Rate Control
- Sinus rhythm (No Intervention)

INTERVENTIONS:
Procedure: Ablation — AV-node ablation
  Arms: AV ablation
Other: Rate Control — Rate control by drug
  Arms: Rate control

SUMMARY:
Examination of CRT efficacy in patients with progressive heart failure and atrial fibrillation at the same time

ELIGIBILITY:
Inclusion Criteria:

* LVEF <35%
* QRS time ≥150ms LBB
* NYHA classification ≥ NYHA III
* permanent (> 6 months) Atrial Fibrillation
* sinus rhythm (control group)
* Condition after Implantation of a Medtronic CRT device
* written informed consent

Exclusion Criteria:

* exchange of the current CRT device
* mitral incompetence (2. degree)
* no compliance
* participation in another study
* pregnancy
* patients with AV node
* patients after heart transplant or those who are on the transplant list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
End systolic left ventricular diameter | 12 months

SECONDARY OUTCOMES:
NYHA-Class, Echo-parameters, ECG-parameters, VO2 max,6 minutes hallwalk-test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Perings, MD, Principal Investigator — marien Hospital Luenen
Locations (1):
- Professor Dr. med. Christian Perings, Lünen, Germany

IPD SHARING:
Plan to Share IPD: No
Not applicable as NO is selected above for 'Plan to share IPD?"